CLINICAL TRIAL: NCT04211714
Title: A Phase I/II Study to Evaluate the Safety and Tolerability of EXG34217 in Patients With Telomere Biology Disorders With Bone Marrow Failure
Brief Title: Study to Evaluate of EXG34217 in Patients With Telomere Biology Disorders With Bone Marrow Failure
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Elixirgen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EXG-US-01
Record Dates: First submitted 2019-12-06; First posted 2019-12-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Telomere Shortening; Bone Marrow Failure
MeSH Terms: conditions — Bone Marrow Failure Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- EXG34217 (Experimental): single autologous CD34+ cells contacted ex vivo with EXG-001
  Interventions: Biological: EXG34217

INTERVENTIONS:
Biological: EXG34217 — Single infusion

SUMMARY:
This is a Phase I/II, open label, single center study to assess the safety and tolerability of EXG34217 in bone marrow failure patients with telomere biology disorders.

DETAILED DESCRIPTION:
This is a Phase I/II, open label study in up to 12 subjects with telomere biology disorders with bone marrow failure. The study is open to all participants regardless of gender or ethnicity. Subjects who are enrolled but not evaluable will be replaced.

Subjects will sign a consent form prior to any study related procedure and will complete baseline screening assessments. Subjects for this study will not require any preparative regimen such as chemotherapy or radiation.

The study will be conducted in three parts

* Peripheral blood mononuclear cells (PBMNCs) collection; mobilization and apheresis,
* Ex vivo cell processing
* Processed cell infusion and post-infusion safety monitoring,
* Follow-up (Week 2, 3,4,5, Months 1, 2,3,4,5,6,9 and 12)

ELIGIBILITY:
Inclusion Criteria:

* Age 12 years and above
* Mild or moderate bone marrow failure defined by satisfying specific conditions.
* Diagnosis of telomere biology disorders

Exclusion Criteria:

* Women of child bearing potential or breastfeeding.
* Patients with cancer who are on active chemotherapeutic treatment.
* Patients with severe bone marrow failure.
* Clonal cytogenetic abnormalities associated with MDS or AML on bone marrow examination.
* Uncontrolled bacterial, viral or fungal infections.
* Prior allogeneic marrow or stem cell transplantation.
* Patients who are not eligible for G-CSF and plerixafor dosing.
* Patients who are not eligible for the apheresis.
* Patients currently taking or have taken danazol and androgens within 60 days prior to Day 1.
* Patients with any other clinically relevant acute or chronic diseases which could interfere with the patients' safety during the trial, expose them to undue risk, or which could interfere with study objectives.
* Patients who have participated in another clinical trial with an investigational drug within the previous 30 days.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2026-10-08 (Estimated); Study Completion 2027-10-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events -Safety by Incidence of Treatment-Emergent Adverse Events | Multiple times for the duration of the study (baseline through Month 12)
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.03. Incidence and nature of adverse events, vital signs, weight.
Number of participants with a change in in physical examination | Multiple times for the duration of the study (baseline through Month 12)
  Physical examination changes General appearance ,Head, eyes, ears, nose, and throat, Respiratory, Cardiovascular, Musculoskeletal, Abdomen, Neurologic, Extremities, Dermatologic, Lymphatic)
Number of participants with a change in Electrocardiography (ECG) | Multiple times for the duration of the study (baseline through Month 12)
  ECG (standard digital 12-lead in singlicate)
Number of participants with a change in clinical laboratory evaluations | Multiple times for the duration of the study (baseline through Month 12)
  Changes in clinical laboratory evaluations (Hematology, Blood chemistry, Coagulation, and Urinalysis)
Number of participants with a change of Immunogenicity | Multiple times for the duration of the study (baseline through Month 12)
  Change in Antibody against virus vector and transgene

SECONDARY OUTCOMES:
Number of participants with a change in telomere length | Screening, Month1,3,6 and 12
  Change in telomere length in any peripheral blood cells
Number of participants with improvement of blood counts. | Multiple times for the duration of the study (baseline through Month 12)
  Blood counts: neutrophils,platelets, or hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Kasiani Myers, MD, Principal Investigator — Cincinnati Children Hospital Medical Center
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Myers KC, Davies SM, Lutzko C, Wahle R, Grier DD, Aubert G, Norris K, Baird DM, Koga M, Ko AC, Amano T, Amano M, Yu H, Ko MSH. Clinical Use of ZSCAN4 for Telomere Elongation in Hematopoietic Stem Cells. NEJM Evid. 2025 Mar;4(3):EVIDoa2400252. doi: 10.1056/EVIDoa2400252. Epub 2025 Feb 25. PMID 39998303